CLINICAL TRIAL: NCT05184283
Title: Longitudinal Assessment of Muscle Health in Patients Undergoing Liver Transplantation (LT) for Hepatocellular Carcinoma (HCC)
Brief Title: Utilization of MAsS in Patients Undergoing LT for HCC
Status: Terminated | Type: Observational
Why Stopped: Discontinued by Amra Medical due to funding.
Sponsor: Columbia University (Other)
Collaborators: Amra Medical AB (Industry)
Responsible Party: Principal Investigator, Julia Wattacheril, Associate Professor of Medicine, Columbia University
Other Study IDs: AAAT7360
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: NAFLD; Hepatocellular Carcinoma; Liver Diseases; Liver Cancer; Cirrhosis, Liver; Hepatitis C
Keywords: NAFLD; Hepatocellular Carcinoma; Liver Diseases; Liver Cancer; Cirrhosis, Liver; Hepatitis C
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Carcinoma, Hepatocellular; Liver Diseases; Liver Neoplasms; Liver Cirrhosis; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: Chart review will be performed for patients who consent to inclusion in the study. Information from routine care will be reviewed and body composition assessment will be done by routine MRI with an additional 6-8 minute scan using AMRA® Profiler 4 Muscle Assessment Score (MAsS) by performing volumetric quantification of fat and water images acquired with 2-point Dixon magnetic resonance imaging (MRI).

SUMMARY:
The aim of this study is to determine the effects of liver transplantation and standard immunosuppression on body composition in patients with compensated cirrhosis and hepatocellular carcinoma.

DETAILED DESCRIPTION:
The combination of hepatocellular carcinoma and chronic liver disease represents a dual impact on overall metabolism. The major risk factors for chronic liver disease related-hepatocellular carcinoma (HCC) include nonalcoholic fatty liver disease (NAFLD), alcoholic liver disease and hepatitis C virus (HCV), among other etiologies of chronic liver injury.

Of particular interest is how the changing landscape of liver disease impacts the care of patients in the peritransplant period. Numerous recent studies have reported that nonalcoholic steatohepatitis (NASH)-related cirrhosis is the most rapidly growing indication for liver transplantation (LT) in the Western world. NAFLD related HCC is already a leading indication in women. The impact of NAFLD on public health and mortality is substantial: incident decompensated cirrhosis due to NAFLD is predicted to increase by 168%, from 39,230 cases annually in 2015 to 105,430 cases in 2030. The corresponding burden of NAFLD cirrhosis on liver transplantation (LT) is expected to increase by 59%. Finally, 3% per year of cirrhotic patients because of NAFLD, develop HCC and noncirrhotic NAFLD-HCC continues to be an area of investigation.

Since NAFLD is becoming one of the most frequent causes of cirrhosis, HCC, and liver transplantation worldwide, it is crucial to identify changes in the peritransplant period that are associated with adverse muscle health and unfavorable metabolic status in the context of all chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Diagnosis of cirrhosis and HCC
* Listed or in evaluation for liver transplantation

Exclusion Criteria:

* History of prior solid organ transplantation
* In evaluation or listed for any other solid organ transplant (other than liver transplant)
* Contraindication to MR examination
* Metastatic HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Undergoing Liver Transplantation for Hepatocellular Carcinoma at risk of nonalcoholic fatty liver disease (NAFLD), alcoholic liver disease and hepatitis C virus (HCV), among other etiologies of chronic liver injury
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Change in mean muscle volume | Baseline (0-12 months prior to transplant), Day 180 (post-transplant), 1 year (post-transplant)
  Muscle volume will be collected using body composition MR image acquisition that adds about 6-8 minutes acquisition time to the clinically prescribed MRI examination.
Change in mean muscle fat | Baseline (0-12 months prior to transplant), Day 180 (post-transplant), 1 year (post-transplant)
  Muscle fat will be collected using body composition MR image acquisition adds about 6-8 minutes acquisition time to the clinically prescribed MRI examination

SECONDARY OUTCOMES:
Survival Rate | Day 90, Day 180, 1 year
  The percentage of people that are still alive at each time point post transplant compare to 89% average survival rate
Number of participants that dropped out of study | 1 year
  This is to measure how many participants did not complete the study for any cause
MRI-proton density fat fraction (MRI-PDFF) | Baseline (0-12 months prior to transplant), Day 180 (post-transplant), 1 year (post-transplant)
  This is to measure/assess intrahepatic fat (IHF) using body composition MR image acquisition adds about 6-8 minutes acquisition time to the clinically prescribed MRI examination
Visceral adipose tissue volume | 1 year
  Visceral adipose tissue volume will be collected using body composition MR image acquisition adds about 6-8 minutes acquisition time to the clinically prescribed MRI examination
Abdominal subcutaneous adipose tissue volume | 1 year
  Abdominal subcutaneous adipose tissue volume will be collected using body composition MR image acquisition adds about 6-8 minutes acquisition time to the clinically prescribed MRI examination
Delta HOMA-IR | 1 year
  Delta homeostasis model assessment of insulin resistance (HOMA-IR) will be assessed using plasma glucose, insulin

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wattacheril, MD, Principal Investigator — Columbia University Irving Medical Center/ New York Presbyterian hospital
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doycheva I, Issa D, Watt KD, Lopez R, Rifai G, Alkhouri N. Nonalcoholic Steatohepatitis is the Most Rapidly Increasing Indication for Liver Transplantation in Young Adults in the United States. J Clin Gastroenterol. 2018 Apr;52(4):339-346. doi: 10.1097/MCG.0000000000000925. PMID 28961576
- [Background] Wong RJ, Aguilar M, Cheung R, Perumpail RB, Harrison SA, Younossi ZM, Ahmed A. Nonalcoholic steatohepatitis is the second leading etiology of liver disease among adults awaiting liver transplantation in the United States. Gastroenterology. 2015 Mar;148(3):547-55. doi: 10.1053/j.gastro.2014.11.039. Epub 2014 Nov 25. PMID 25461851
- [Background] Cholankeril G, Wong RJ, Hu M, Perumpail RB, Yoo ER, Puri P, Younossi ZM, Harrison SA, Ahmed A. Liver Transplantation for Nonalcoholic Steatohepatitis in the US: Temporal Trends and Outcomes. Dig Dis Sci. 2017 Oct;62(10):2915-2922. doi: 10.1007/s10620-017-4684-x. Epub 2017 Jul 25. PMID 28744836
- [Background] Parikh ND, Marrero WJ, Wang J, Steuer J, Tapper EB, Konerman M, Singal AG, Hutton DW, Byon E, Lavieri MS. Projected increase in obesity and non-alcoholic-steatohepatitis-related liver transplantation waitlist additions in the United States. Hepatology. 2019 Aug;70(2):487-495. doi: 10.1002/hep.29473. Epub 2018 May 14. PMID 28833326
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Linge J, Borga M, West J, Tuthill T, Miller MR, Dumitriu A, Thomas EL, Romu T, Tunon P, Bell JD, Dahlqvist Leinhard O. Body Composition Profiling in the UK Biobank Imaging Study. Obesity (Silver Spring). 2018 Nov;26(11):1785-1795. doi: 10.1002/oby.22210. Epub 2018 May 22. PMID 29785727
- [Background] Linge J, Ekstedt M, Dahlqvist Leinhard O. Adverse muscle composition is linked to poor functional performance and metabolic comorbidities in NAFLD. JHEP Rep. 2020 Oct 28;3(1):100197. doi: 10.1016/j.jhepr.2020.100197. eCollection 2021 Feb. PMID 33598647
- [Background] Linge J, Heymsfield SB, Dahlqvist Leinhard O. On the Definition of Sarcopenia in the Presence of Aging and Obesity-Initial Results from UK Biobank. J Gerontol A Biol Sci Med Sci. 2020 Jun 18;75(7):1309-1316. doi: 10.1093/gerona/glz229. PMID 31642894
- [Background] Borga M, Thomas EL, Romu T, Rosander J, Fitzpatrick J, Dahlqvist Leinhard O, Bell JD. Validation of a fast method for quantification of intra-abdominal and subcutaneous adipose tissue for large-scale human studies. NMR Biomed. 2015 Dec;28(12):1747-53. doi: 10.1002/nbm.3432. Epub 2015 Nov 2. PMID 26768490
- [Background] West J, Romu T, Thorell S, Lindblom H, Berin E, Holm AS, Astrand LL, Karlsson A, Borga M, Hammar M, Leinhard OD. Precision of MRI-based body composition measurements of postmenopausal women. PLoS One. 2018 Feb 7;13(2):e0192495. doi: 10.1371/journal.pone.0192495. eCollection 2018. PMID 29415060
- [Background] West J, Dahlqvist Leinhard O, Romu T, Collins R, Garratt S, Bell JD, Borga M, Thomas L. Feasibility of MR-Based Body Composition Analysis in Large Scale Population Studies. PLoS One. 2016 Sep 23;11(9):e0163332. doi: 10.1371/journal.pone.0163332. eCollection 2016. PMID 27662190
- [Background] Karlsson A, Rosander J, Romu T, Tallberg J, Gronqvist A, Borga M, Dahlqvist Leinhard O. Automatic and quantitative assessment of regional muscle volume by multi-atlas segmentation using whole-body water-fat MRI. J Magn Reson Imaging. 2015 Jun;41(6):1558-69. doi: 10.1002/jmri.24726. Epub 2014 Aug 11. PMID 25111561
- [Background] Ajmera VH, Cachay E, Ramers C, Vodkin I, Bassirian S, Singh S, Mangla N, Bettencourt R, Aldous JL, Park D, Lee D, Blanchard J, Mamidipalli A, Boehringer A, Aslam S, Leinhard OD, Richards L, Sirlin C, Loomba R. MRI Assessment of Treatment Response in HIV-associated NAFLD: A Randomized Trial of a Stearoyl-Coenzyme-A-Desaturase-1 Inhibitor (ARRIVE Trial). Hepatology. 2019 Nov;70(5):1531-1545. doi: 10.1002/hep.30674. Epub 2019 Jun 18. PMID 31013363
- [Background] Middleton MS, Haufe W, Hooker J, Borga M, Dahlqvist Leinhard O, Romu T, Tunon P, Hamilton G, Wolfson T, Gamst A, Loomba R, Sirlin CB. Quantifying Abdominal Adipose Tissue and Thigh Muscle Volume and Hepatic Proton Density Fat Fraction: Repeatability and Accuracy of an MR Imaging-based, Semiautomated Analysis Method. Radiology. 2017 May;283(2):438-449. doi: 10.1148/radiol.2017160606. Epub 2017 Mar 9. PMID 28278002